CLINICAL TRIAL: NCT04933253
Title: Mediastinal Temperature and Post-operative Bleeding
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment has been unsuccessful and the study team is withdrawing the study while they consider options and alternatives.
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HM20021183
Record Dates: First submitted 2021-06-14; First posted 2021-06-21 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Blood Loss, Surgical
MeSH Terms: conditions — Blood Loss, Surgical

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): this cohort will receive 2 L of warm 37celsius saline irrigation of the mediastinum prior to closure of the chest
  Interventions: Procedure: Saline irrigation
- Control (No Intervention): this cohort will receive the normal standard of care as established by the primary surgeon

INTERVENTIONS:
Procedure: Saline irrigation — Mediastinal irrigation with 2 L of 37 degree Celsius saline prior to chest closure
  Arms: Experimental

SUMMARY:
This study will investigate how chest temperature relates to blood loss and blood clotting. Researchers will use infra-red thermometers to measure the temperature of the chest at the end of surgery see if this relates to the amount of blood collected from the surgical drains. In addition, researchers will test if warm irrigation of the chest increases the temperature of the chest and if this impacts blood loss.

DETAILED DESCRIPTION:
Low body temperature during surgery, defined as a temperature below 34 °C, occurs commonly in patients undergoing cardiac surgery due to the bypass machine and an open chest. Low body temperature has been associated with blood loss, but the relevant published data are inconclusive. Nevertheless, evidence suggests that blood loss during and after surgery are higher in low body temperature patients than in the normal body temperature patients. In addition, low body temperature can impair blood clotting. The clinical significance of this is high as it is well established that blood transfusion increases mortality after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing open cardiac surgery at VCU
* Age18 to 80 years
* American Society of Anesthesiologists Physical Status 1-3

Exclusion Criteria:

* history of excessive bleeding
* partial thromboplastin time > 35 s
* prothrombin time > 35 s
* fibrinogen < 200 mg/dL
* platelet count < 100,000/L
* history of infection and fever within 4 weeks before surgery
* use of steroid or immunosuppressant within 4 weeks before surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Chest temperature | At the end of surgery, up to 5 hours
  We will use infra-red thermometers to measure the temperature of the chest at the end of surgery
Amount of blood loss | 24 hours after the end of surgery
  amount of blood drained into the cell-saving device or collection canisters from the chest drains that are left in all patients after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Arturo Cardounel, M.D., Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No